CLINICAL TRIAL: NCT01495780
Title: Feasibility and Cost Effectiveness of Physiological Monitoring at Home in COPD Patients
Brief Title: eRT Remote Health Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: eResearch Technology (eRT) (Unknown)
Responsible Party: Principal Investigator, Christopher B Cooper, MD, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: eRT RHM
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; COPD; Chronic Obstructive Lung Disease; Bronchitis, Chronic; Pulmonary Emphysema
Keywords: Behavioral; Remote monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Pulmonary Emphysema; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remote Health Monitoring (Experimental): Subjects assigned to this arm will conduct daily at-home health monitoring using several electronic devices that will transmit data back to the study team. Everyday, subjects will measure pulse oximetry (SpO2) using a finger clip, answer questions about symptoms and medication use, answer a quality of life questionnaire, perform breathing tests, and record physical activity (using a physical activity monitor that will be mailed to the study team). Wearing the activity monitor is optional and will only occur during months 1, 6, and 12.
  Interventions: Behavioral: Remote Health Monitoring

INTERVENTIONS:
Behavioral: Remote Health Monitoring — 1 year of remote health monitoring of symptoms, medication use, breathing tests, physical activity, and healthcare utilization.

SUMMARY:
Remote Health Monitoring (RHM) is the assessment of one's own symptoms at home between doctor visits, using things like at-home breathing tests, electronic diaries to answer questionnaires, and other monitoring devices. The hypothesis of this study is that the health and quality of life of people with COPD who do RHM for one year will be better than people with COPD who do not do RHM. Subjects who are at least 40 years old, have been diagnosed with chronic obstructive pulmonary disease (COPD), also known as chronic bronchitis or emphysema, and are current or former smokers will be invited to participate. This study is paid for by eResearch Technology (eRT).

Subjects will complete 2 visits at UCLA, separated by one year of RHM. All subjects will participate in RHM. RHM will involve daily monitoring at home using a few electronic devices: blood oxygen levels, symptoms, medication use, breathing tests, and activity monitoring. Visits will include physical exam and medical history, ECG, questionnaires, breathing tests, and exercise tests.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years.
* Clinical diagnosis of moderate to severe COPD in accordance with the definition of the American Thoracic Society (ATS).9
* Smoking history >10 pack-years.
* Postbronchodilator FEV1/FVC<70% and FEV1<70% based on NHANES III reference values
* Domestic situation felt to be supportive of remote health monitoring.
* Ability to give informed consent.

Exclusion Criteria:

* Clinical diagnosis of asthma.
* Pulmonary disease other than COPD (e.g., lung cancer, sarcoidosis, active tuberculosis, bronchiectasis, pulmonary fibrosis, cystic fibrosis, or alpha-1-antitrypsin deficiency) or had lung volume reduction.
* Any other active disease that, in the opinion of the investigator, would put the safety of the subject at risk through study participation (e.g. unstable cardiovascular disease, renal failure, stroke).
* Previously diagnosed cancer is considered a significant disease unless it is in complete remission for 2 years at the initial visit.
* Any other disease that is life-threatening and carries a prognosis less than two years that, in the opinion of the investigator, is likely to influence the clinical course during the conduct of this trial.
* Myocardial infarction within 6 weeks of enrolment.
* Use of long-term oxygen therapy (LTOT) prescribed for greater than 12 hours a day.
* A known or suspected history of drug or alcohol abuse within 2 years prior to the initial visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-08-20 (Actual); Study Completion 2014-08-20 (Actual)

PRIMARY OUTCOMES:
Compliance with daily RHM | 1 year
  Compliance with daily RHM as a percentage of study days
Integrity of spirometric data | 1 year
  Integrity of the spirometric data in terms of the standard American Thoracic Society and European Respiratory Society criteria for acceptability and repeatability.

SECONDARY OUTCOMES:
Rate of adoption of RHM | 1 year
  Time it takes for subjects to become compliant with daily RHM
Treatment adherence | 1 year
  Treatment adherence in terms of percentage of days prescribed treatment* is taken (* treatment separate from study, prescribed by personal physician)
Time to first COPD exacerbation | 1 year
  Time to first COPD exacerbation as defined by standard criteria.
Number of COPD exacerbations per year | 1 year
Proportion of subjects experiencing one or more exacerbations | 1 year
Mean daily FEV1 | 1 year
Mean daily IC | 1 year
Mean daily activity level | 1 year
Mean daily SpO2 | 1 year
Daily symptom scores | 1 year
Number of physician visits | 1 year
Number of emergency department visits | 1 year
Number of hospitalizations | 1 year
Number of days spent in hospital | 1 year
Health care costs | 1 year
  Inferred health care costs using a standard cost framework model

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Cooper, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Los Angeles, California, United States